CLINICAL TRIAL: NCT02636556
Title: Phase Ⅱ Study of Concurrent Chemoradiotherapy for Limited Advanced Unresectable Thymic Epithelial Tumors
Brief Title: Chemoradiotherapy for Limited Advanced Unresectable Thymic Epithelial Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kailiang Wu, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508151-5
Record Dates: First submitted 2015-12-15; First posted 2015-12-21 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Thymoma and Thymic Carcinoma
Keywords: thymoma; thymic carcinoma; chemoradiotherapy; inoperable
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Intervention Model Description: Intensity modulated radiotherapy with VP-16/Cisplatin
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemoradiation (Experimental): concurrent chemoradiation.
  Interventions: Radiation: concurrent chemoradiation

INTERVENTIONS:
Radiation: concurrent chemoradiation — The patients receive chemotherapy concurrent with Radiotherapy. The prescription dose is 60Gy in 30 fractions in 6 weeks.The chemotherapy regimen is cisplatin (25mg/m2,iv drip,d1-3) and etoposide (75mg/m2,iv drip,d1-3),q4w*4.

SUMMARY:
This study is designed to evaluate the feasibility and safety of concurrent chemoradiotherapy for limited advanced unresectable thymoma or thymic carcinoma.

DETAILED DESCRIPTION:
Complete resection is difficult to achieve without damaging the main organs in advanced thymoma or thymic carcinoma. The previous trials have showed that radiotherapy was significantly associated with prolonged OS and chemotherapy is playing an increasing role in treatment of patients with advanced thymoma or thymic carcinoma. However, whether concurrent chemoradiotherapy is safety in advanced thymoma or thymic carcinoma is still unknown. The purpose of this study is to evaluate the feasibility and safety of concurrent chemoradiotherapy for limited advanced unresectable thymoma or thymic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1.18~75 years old; 2.Eastern Cooperative Oncology Group performance status of 0 to 2; 3.Pathologically or cytologically confirmed untreated thymoma or thymic carcinoma; 4.Unresectable, limited adanced disease could be encompassed within a tolerable radiotherapy field; 5.Have adequate bone marrow, hepatic, and renal function; 6.Patients who cannot receive surgery resection; 7.Written informed consent.

Exclusion Criteria:

1. Distant metastases could not be encompassed within a tolerable radiotherapy field;
2. Underwent surgery, radiotherapy or chemotherapy before entering this study ;
3. Have other malignancy history excluding carcinoma in situ of cervix in the previous five years;
4. Active clinical pulmonary infection;
5. Pregnant or nursing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 3 months after treatment
  Evaluated using RECIST (Response Evaluation Criteria in Solid Tumors) 1.0 criteria

SECONDARY OUTCOMES:
Overall survival | 2 years
  from registration to death as a result of any cause.
Progression free survival | 2 years
  from registration to first documentation of disease progression or death.
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v4.0 | up to 2 years
  Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Kailiang Wu, M.D.,Ph.D, Principal Investigator — Fudan University
Locations (1):
- Kailiang Wu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No